CLINICAL TRIAL: NCT05018403
Title: A Randomized, Single-center, Double-blind, Placebo Controlled, First-in-human Trial With Single Ascending Intravenous Doses to Determine Safety, Tolerability and Pharmacokinetics of AON-D21 in Healthy Male Subjects
Brief Title: First-in-human Trial With Single-dose C5a-neutralizing AON-D21 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptarion Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-D21-C100; 2021-000935-30 (EudraCT Number)
Record Dates: First submitted 2021-08-10; First posted 2021-08-24 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Five groups of participants will be assigned to receive AON-D21 or placebo in ascending dose order. Doses will be escalated based on safety and pharmacokinetic data.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple: Participant, Investigator, Outcomes Assessor and Care provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AON-D21 (Experimental): Single ascending doses by iv infusion.
  Interventions: Drug: Intravenous AON-D21
- Placebo (Placebo Comparator): Placebo medication identical in appearance to active.
  Interventions: Drug: Intravenous placebo

INTERVENTIONS:
Drug: Intravenous AON-D21 — AON-D21 is a Pegylated L-configured aptamer that binds and thereby neutralizes the complement component C5a from activating both C5a receptors.
  Other Names: AON-D21
  Arms: AON-D21
Drug: Intravenous placebo — Isotonic glucose solution identical in appearance to AON-D21.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamic parameters after single ascending intravenous doses of AON-D21 in healthy male subjects.

DETAILED DESCRIPTION:
This study will potentially include 5 sequential cohorts with 8 subjects per cohort, then 40 enrolled subjects in total. Within each dose group 6 subjects will be randomized to receive AON-D21 and 2 subjects will be randomly assigned to placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Body mass index (BMI) within the range 18 - 30 kg/m2 with a body weight between 50 kg and 120 kg.
* Male subjects
* Subject is healthy as determined by medical evaluation
* Subject provided written informed consent
* Subject is willing to comply with all requirements and restrictions according to the study protocol.

Exclusion Criteria:

* Any concomitant disease, condition, or treatment that could interfere with the conduct of the study.
* Any acquired or congenital immune deficiency.
* Acute infection (including viral infections) in the preceding 6 weeks (8 weeks for respiratory infections).
* Any concomitant disease, condition, or treatment that could interfere with the conduct of the study.
* Any acquired or congenital immune deficiency.
* Acute infection (including viral infections) in the preceding 6 weeks (8 weeks for respiratory infections).
* Clinically relevant abnormality following the Investigator's review of the physical examination, vital signs, ECG and clinical study protocol-defined clinical laboratory tests that, in the opinion of the Investigator, would preclude inclusion in the trial at screening and admission.
* Evidence of COVID-19 signs or symptoms, exposure to infected person or confirmed COVID-19 infection within the last 2 weeks.
* Use of any concomitant medication or prescribed or non-prescribed drugs within 2 weeks or 5 times the half-life, whichever is longer, prior to the first study treatment administration.
* Administration of vaccine(s) within 2 weeks prior to screening or plans to receive such vaccines during the study.
* Use of any investigational drug or participation in any clinical study within 30 days or 5 half-life times, whichever is longer, prior to dosing.
* Positive drug or alcohol screen at screening and admission.
* Any significant blood loss, donated one unit (450 mL) of blood or more, or donated plasma, or received a transfusion of any blood or blood products within 30 days prior to dosing.
* Subjects who are unable to refrain from the consumption of Seville oranges, grapefruit or grapefruit juice and /or pomelos, exotic citrus fruits, grapefruit hybrids, starfruit or fruit juices from 72 hours prior to dosing on Day 1, until completion of the last pharmacokinetic (PK) blood sample time point.
* Legal incapacity or limited legal capacity, or incarceration.
* Inability to understand or communicate reliably with the Investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Overall number of participants with treatment-emergent adverse events (TEAEs) per dosing cohort as assessed by CTCAE. | 14 days.
  To determine the overall safety and tolerability of AON-D21 by analyzing number of participants with treatment-related adverse events as assessed by CTCAE. Nature, occurrence, and severity of treatment-emergent adverse events.
Primary Safety Endpoint - Per Dosing Cohort number of participants with treatment-emergent adverse events as assessed by CTCAE. | 14 days
  Overall number of participants with treatment related treatment-emergent adverse events (TEAEs) as assessed by CTCAE per dosing cohort.

SECONDARY OUTCOMES:
Pharmacokinetics of AON-D21. | 14 days.
  To determine the area under the concentration (AUC)-time curve from 0 to 48 h (AUC0-48).
Pharmacokinetics of AON-D21. | 14 days.
  To determine the area under the concentration (AUC)-time curve from 0 to 72 h (AUC0-72).
Pharmacokinetics of AON-D21. | 14 days.
  To determine the area under the concentration (AUC)-time curve from 0 to infinity (AUC0-inf).
Pharmacokinetics of AON-D21. | 14 days.
  To determine the maximum concentration (Cmax).
Pharmacokinetics of AON-D21. | 14 days.
  To determine the time of maximum concentration (Tmax).
Pharmacokinetics of AON-D21. | 14 days.
  To determine the half-life (t1/2).
Pharmacokinetics of AON-D21. | 14 days.
  To determine the plasma clearance (CL) calculated as Dose/AUC0-inf.
Pharmacokinetics of AON-D21. | 14 days.
  To determine the volume of distribution (Vz).
Pharmacokinetics of AON-D21. | 14 days.
  To determine the amount of AON-D21 excreted (Ae) in urine.
Pharmacokinetics of AON-D21. | 14 days.
  To determine the renal clearance (CLR) of AON-D21.

OTHER OUTCOMES:
Pharmacodynamics | 14 days
  To determine the C5a inhibition capacity of AON-D21 by measuring active C5a in blood using a cell-based assay.
Effects on the complement status | 14 days
  Determining the effect of AON-D21 on levels of C5, C5a, C5b-9 in blood and on the capacity of terminal complement complex formation.
To assess potential for immunogenicity of AON-D21 | 14 days
  Determining the presence of anti-drug antibodies (ADA) and anti-peg antibodies in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Koch, MD, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No